CLINICAL TRIAL: NCT06719986
Title: A Study to Characterize the Time Course of Reversal of Opioid (Fentanyl)-Induced Respiratory Depression Following Administration of Nalmefene Autoinjector 1.5 mg (0.94% MgCl2) Intramuscular and Narcan® 4 mg Intranasal in Healthy Subjects
Brief Title: Pharmacodynamic Evaluation of Intramuscular Nalmefene Autoinjector 1.5 mg Compared to Intranasal Narcan 4 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NAL1004
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose | interventions — nalmefene; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nalmefene Hydrochloride (HCl) injection (Experimental): Nalmefene Hydrochloride injection 1.5 mg for intramuscular (IM) administration
  Interventions: Drug: Nalmefene HCl injection
- Narcan intranasal (Active Comparator): Naloxone 4 mg for intranasal (IN) administration
  Interventions: Drug: Naloxone HCl intranasal

INTERVENTIONS:
Drug: Nalmefene HCl injection — Nalmefene Hydrochloride injection 1.5 mg for intramuscular (IM) administration
  Arms: Nalmefene Hydrochloride (HCl) injection
Drug: Naloxone HCl intranasal — Naloxone 4 mg for intranasal (IN) administration
  Other Names: Narcan
  Arms: Narcan intranasal

SUMMARY:
The purpose of this study is to determine the pharmacodynamics (change in minute ventilation) of nalmefene when given as an autoinjector intramuscularly (IM; into the thigh) compared to naloxone when given intranasally (IN; into the nose) to healthy subjects with prior opioid exposure under steady state fentanyl concentrations (opioid agonism).

ELIGIBILITY:
Key Inclusion Criteria include:

1. Healthy and free of significant abnormal findings as determined by medical history, physical examination, clinical laboratory values, vital signs, and ECG.
2. Body weight ranging from 50 to 100 kg (110-220 lbs) and body mass index (BMI) within the range [18-30] kg/m2 (inclusive).
3. Willing to be compliant with the protocol, capable of subjective evaluation, if applicable, able to read and understand questionnaires, if applicable.

Key Exclusion Criteria include:

1. Females who are pregnant or lactating.
2. Any significant illness during the 30 days preceding the initial dose in this study.
3. History or any current conditions that might interfere with drug absorption, distribution, metabolism or excretion.
4. Refusal to abstain from caffeine or xanthine containing beverages entirely during confinement.
5. Refusal to abstain from consumption of alcoholic beverages 48 hours prior to initial study drug administration and through the end-of-study visit.
6. Difficulty with venous access or unsuitable for or unwilling to undergo catheter insertion.

Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio Clinical Trials, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was dosed 03-October-2022 and the last subject completed the study 23-December-2022. The study was conducted at 1 site in the US.
Pre-assignment Details: The Qualification Phase (Part 1) was conducted prior to the Treatment Phase (Part 2) to identify subjects eligible for participation in Part 2. N=13 subjects who had not previously qualified in a similar study at the same site and N=11 subjects who had previously qualified in a similar study at the same site for a total of N=24 subjects who participated in the Treatment Phase (Part 2).
Groups:
- Fentanyl Infusion: The Qualification Phase (Part 1) was conducted prior to Part 2 to identify subjects who had not previously qualified in a similar study at the same site. During Qualification, subjects were given an IV infusion of fentanyl titrated to produce up to an average of 50% decrease in minute ventilation.
- Sequence 1 (Test-Reference-Test-Reference): Treatment Phase (Part 2) - Sequence 1 - BABA.
  This was a 4-period, 2-treatment, 2-sequence, replicate randomization.
  Subjects received a single dose of Nalmefene Hydrochloride injection 1.5 mg for IM administration (Treatment B [Test]) on Day 1 in Period 1, then a single dose of Naloxone 4 mg for IN administration (Treatment A [Reference] on Day 1 in Period 2, then a single dose of Nalmefene Hydrochloride injection 1.5 mg for IM administration (Treatment B [Test]) on Day 1 in Period 3, then a single dose of Naloxone 4 mg for IN administration (Treatment A [Reference] on Day 1 in Period 4.
  All completed subjects received two rounds of Nalmefene and 2 rounds of Naloxone.
- Sequence 2 (Reference-Test-Reference-Test): Treatment Phase (Part 2) - Sequence 2 - ABAB.
  This was a 4-period, 2-treatment, 2-sequence, replicate randomization.
  Subjects received a single dose of Naloxone 4 mg for IN administration (Treatment A [Reference]) on Day 1 in Period 1, then a single dose of Nalmefene Hydrochloride injection 1.5 mg for IM administration (Treatment B [Test]) on Day 1 in Period 2, then a single dose of Naloxone 4 mg for IN administration (Treatment A [Reference]) on Day 1 in Period 3, then a single dose of Nalmefene Hydrochloride injection 1.5 mg for IM administration (Treatment B [Test]) on Day 1 in Period 4.
  All completed subjects received two rounds of Naloxone and 2 rounds of Nalmefene.
Period: Part 1 Qualification (1 Day)
Arm/Group | Fentanyl Infusion | Sequence 1 (Test-Reference-Test-Reference) | Sequence 2 (Reference-Test-Reference-Test)
Started | 13 | 0 | 0
Completed | 13 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Qualification Washout (12 Hours)
Arm/Group | Fentanyl Infusion | Sequence 1 (Test-Reference-Test-Reference) | Sequence 2 (Reference-Test-Reference-Test)
Started | 13 | 0 | 0
Completed | 13 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part 2 Period 1 (1 Day)
Arm/Group | Fentanyl Infusion | Sequence 1 (Test-Reference-Test-Reference) | Sequence 2 (Reference-Test-Reference-Test)
Started (13 subjects qualified for Part 2 in the Qualification Phase (Part 1) and 11 subjects previously qualified for Part 2 in a similar study at the same site.) | 0 | 12 | 12
Completed | 0 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Washout (up to 72 Hours)
Arm/Group | Fentanyl Infusion | Sequence 1 (Test-Reference-Test-Reference) | Sequence 2 (Reference-Test-Reference-Test)
Started | 0 | 12 | 12
Completed | 0 | 12 | 11
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Period: Part 2 Period 2 (1 Day)
Arm/Group | Fentanyl Infusion | Sequence 1 (Test-Reference-Test-Reference) | Sequence 2 (Reference-Test-Reference-Test)
Started | 0 | 12 | 11
Completed | 0 | 12 | 11
Not Completed | 0 | 0 | 0
Period: Washout (up to 72 Hours)
Arm/Group | Fentanyl Infusion | Sequence 1 (Test-Reference-Test-Reference) | Sequence 2 (Reference-Test-Reference-Test)
Started | 0 | 12 | 11
Completed | 0 | 12 | 11
Not Completed | 0 | 0 | 0
Period: Part 2 Period 3 (1 Day)
Arm/Group | Fentanyl Infusion | Sequence 1 (Test-Reference-Test-Reference) | Sequence 2 (Reference-Test-Reference-Test)
Started | 0 | 12 | 11
Completed | 0 | 12 | 11
Not Completed | 0 | 0 | 0
Period: Washout (up to 72 Hours)
Arm/Group | Fentanyl Infusion | Sequence 1 (Test-Reference-Test-Reference) | Sequence 2 (Reference-Test-Reference-Test)
Started | 0 | 12 | 11
Completed | 0 | 11 | 11
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Part 2 Period 4 (1 Day)
Arm/Group | Fentanyl Infusion | Sequence 1 (Test-Reference-Test-Reference) | Sequence 2 (Reference-Test-Reference-Test)
Started | 0 | 11 | 11
Completed | 0 | 11 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Subjects received Nalmefene Hydrochloride injection 1.5 mg for intramuscular (IM) administration or Naloxone 4 mg for intranasal (IN) administration in a crossover fashion according to the randomization sequence.
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (7.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 10
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Minute Ventilation 5 Minutes From Opioid Induced Nadir
Description: To assess the change in minute ventilation at 5 minutes of intramuscular nalmefene and intranasal naloxone reversal from the opioid induced nadir.
Time Frame: 5 minutes after opioid antagonist administration
Population: Eligible analysis set was defined as subjects/periods who were randomized, received study drug, had at least 1 valid pharmacodynamic (PD) measurement, and their opioid-induced respiratory depressions (OIRDs) were worse than baseline for minute ventilation (MV) and transcutaneous CO2 (TCO2). The data for the overall treatment period was calculated as the average of available data from individual periods.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 24
L/min | 4.42 (2.033) | 2.03 (0.992)

2. Secondary Outcome: Change in Minute Ventilation at 2.5, 5, 10, 15, 20, 30, and 90 Minutes From Opioid Induced Nadir
Description: To assess the time course of changes in minute ventilation of intramuscular nalmefene and intranasal naloxone reversal from the opioid induced nadir.
Time Frame: Baseline, 2.5, 5, 10, 15, 20, 30, and 90 minutes after opioid antagonist administration
Population: Eligible analysis set was defined as subjects/periods who were randomized, received study drug, had at least 1 valid pharmacodynamic (PD) measurement, and their opioid-induced respiratory depressions (OIRDs) were worse than baseline for minute ventilation (MV) and transcutaneous CO2 (TCO2). The data for overall treatment period was calculated as the average of available data from individual periods.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 24
L/min
  Baseline | 2.92 (1.254) | 3.02 (1.022)
  2.5 minutes | 2.00 (1.284) | 1.67 (1.046)
  5 minutes | 4.42 (2.033) | 2.03 (0.992)
  10 minutes | 3.97 (1.755) | 2.57 (1.364)
  15 minutes | 4.15 (1.990) | 2.79 (1.328)
  20 minutes | 4.00 (2.176) | 3.11 (1.160)
  30 minutes | 3.62 (1.820) | 2.92 (1.357)
  90 minutes | 2.74 (1.519) | 2.55 (0.994)

3. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum plasma concentration of nalmefene and naloxone.
Time Frame: up to 24 hours post-dose
Population: Full analysis population was defined as all subjects who were randomized, received study drug and had at least 1 valid pharmacodynamics (PD) measurement. Pharmacokinetic analyses and summaries were based on the full analysis population. For the overall analysis, the values were averaged within each subject first, then the descriptive statistics were calculated.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 24
ng/mL | 8.3576 (3.71139) | 5.6015 (2.30753)

4. Secondary Outcome: Area Under the Curve (AUC0-2.5)
Description: Area under the plasma concentration-time curve from time zero to 2.5 minutes
Time Frame: 2.5 minutes post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 24
ng*hr/mL | 0.0440 (0.03923) | 0.256 (0.03663)

5. Secondary Outcome: Area Under the Curve (AUC0-5)
Description: Area under the plasma concentration-time curve from time zero to 5 minutes
Time Frame: 5 minutes post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 24
ng*hr/mL | 0.2225 (0.13565) | 0.1002 (0.11542)

6. Secondary Outcome: Area Under the Curve (AUC0-10)
Description: Area under the plasma concentration-time curve from time zero to 10 minutes
Time Frame: 10 minutes post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 24
ng*hr/mL | 0.7576 (0.38147) | 0.3311 (0.27201)

7. Secondary Outcome: Area Under the Curve (AUC0-15)
Description: Area under the plasma concentration-time curve from time zero to 15 minutes
Time Frame: 15 minutes post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 24
ng*hr/mL | 1.2716 (0.52366) | 0.6300 (0.43256)

8. Secondary Outcome: Area Under the Curve (AUC0-20)
Description: Area under the plasma concentration-time curve from time zero to 20 minutes
Time Frame: 20 minutes post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 24
ng*hr/mL | 1.7479 (0.61346) | 0.9817 (0.61050)

9. Secondary Outcome: Area Under the Curve (AUCt)
Description: Area under the plasma concentration-time curve from time zero to the time of last measurable concentration.
Time Frame: up to 24 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 23
ng*hr/mL | 23.1620 (3.60968) | 13.4803 (2.78735)

10. Secondary Outcome: Area Under the Curve (AUCinf)
Description: Area under the plasma concentration-time curve from time zero to infinity.
Time Frame: up to 24 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 22
ng*hr/mL | 25.7412 (4.65028) | 13.4938 (2.87023)

11. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time to maximum plasma concentration of nalmefene and naloxone.
Time Frame: up to 24 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 24
hour | 0.2083 [0.062 to 1.017] | 0.6667 [0.167 to 1.000]

12. Secondary Outcome: Time to First Measurable Plasma Concentration (Tlag)
Description: Time to first measurable plasma concentration of nalmefene and naloxone.
Time Frame: up to 24 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 24
hour | 0.0527 (0.01912) | 0.0464 (0.01023)

13. Secondary Outcome: Half-life (T1/2)
Description: Half life of nalmefene and naloxone.
Time Frame: up to 24 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
Number analyzed (Participants) | 23 | 22
hour | 7.9754 (2.16550) | 1.6353 (.050257)

ADVERSE EVENTS:
Time Frame: All serious adverse events and adverse events were collected from the signing of the informed consent for study participation through 30 days after the subject's last dose of study drug or within 30 days after the last study visit or follow-up phone call (up to approximately 78 days).
Arm/Group | Fentanyl Infusion | Nalmefene Hydrochloride (HCl) Injection | Narcan Intranasal
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 9/13 | 20/23 | 18/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl Infusion (N=13) | Nalmefene Hydrochloride (HCl) Injection (N=23) | Narcan Intranasal (N=24)
Palpitations (Cardiac disorders) | 0 | 4 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 4 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2
Vomitting (Gastrointestinal disorders) | 0 | 3 | 1
Feeling hot (General disorders) | 1 | 11 | 4
Chills (General disorders) | 0 | 6 | 0
Feeling abnormal (General disorders) | 0 | 3 | 0
Feeling cold (General disorders) | 0 | 2 | 1
Injection site pain (General disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 5 | 5
Dysgeusia (Nervous system disorders) | 0 | 1 | 7
Allodynia (Nervous system disorders) | 0 | 5 | 2
Dizziness (Nervous system disorders) | 2 | 4 | 1
Burning sensation (Nervous system disorders) | 0 | 3 | 0
Irritability (Psychiatric disorders) | 0 | 3 | 1
Agitation (Psychiatric disorders) | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 3
Hot flush (Vascular disorders) | 1 | 3 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0 | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT06719986/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT06719986/SAP_001.pdf